CLINICAL TRIAL: NCT05064501
Title: Impact of COVID19 on Lung Function and Control of Asthma Patients
Brief Title: Impact of COVID19 on Asthma Patients in Spain
Acronym: IMCAS
Status: Withdrawn | Type: Observational
Why Stopped: Difficulty in recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-129
Record Dates: First submitted 2021-09-30; First posted 2021-10-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2022-08

CONDITIONS: Asthma; Covid19
Keywords: asthma; asthma control; COVID19
MeSH Terms: conditions — Asthma; COVID-19 | interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma and COVID19 infection: Asthma and COVID19 infection
  Interventions: Diagnostic Test: spirometry; Other: Asthma control test
- Asthma without COVID19 infection: Asthma and COVID19 infection
  Interventions: Diagnostic Test: spirometry; Other: Asthma control test

INTERVENTIONS:
Diagnostic Test: spirometry — Lung function test: pre and post bronchodilator spirometry
Other: Asthma control test — Asthma control test

SUMMARY:
This research project aims to investigate the impact of COVID-19 on asthmatic patients, particularly focusing on whether the viral infection exacerbates asthma or affects control and lung function in the short to medium term. The study plans to collect and compare data from two groups of asthmatic individuals - those who have experienced a SARS-CoV-2 infection requiring emergency consultation or hospitalization and a matched control group without such infection. Both groups will be followed for one year, with lung function tests conducted at six months and monitoring of exacerbations and changes in Asthma Control Test (ACT) throughout the year. The objective is to enhance understanding of how COVID-19 affects asthmatic patients, leading to improved recommendations, preventive measures, and treatment adjustments based on the study's findings.

DETAILED DESCRIPTION:
The COVID19 pandemic is having an immeasurable impact on the economy and on morbidity and mortality. Knowledge and scientific evidence about this disease is advancing rapidly, but it is not yet known whether asthmatic patients suffering from COVID19 have an exacerbation of asthma, or whether this viral infection has an impact on control and lung function in the short to medium term.

The aim of this study is to define the changes that occur in these two parameters in asthmatic patients suffering from COVID19. To this end, asthmatic patients who have suffered a SARS-CoV-2 infection and who have required an emergency consultation or hospitalisation will be collected in a pneumology consultation and matched by age, sex and severity of asthma with a group that has not suffered the same. Both will be followed for one year, and lung function will be tested at six months and exacerbations and changes in ACT during the following year.

These data are intended to improve the available knowledge on the impact of IDVC19 on asthma patients with a view to making appropriate recommendations, prevention and treatment adjustments in line with the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* 12 -80 years
* Asthma diagnosis according to guidelines
* Follow up on asthma clinics in one of the participant hospitals

Exclusion Criteria:

* Other severe respiratory condition independent of asthma

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients between the ages of 12 and 80 diagnosed with asthma according to current guidelines (GEMA/GINA), of any level of severity, will be recruited and followed up in Pneumology consultations at participating hospitals. The study cohort would be patients with these criteria who have needed to consult the Emergency Department or be admitted for COVID19 (suggestive symptomatology + CRP and/or positive serology) in the six months prior to the visit. The control group would be a cohort of asthmatic patients matched by age, severity and sex, who have not suffered COVID19 or compatible symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Asthma control | 6 months
  Change in score of Asthma Control Test (ACT). Min 5 máx 25 (the higher score indicates better control)

SECONDARY OUTCOMES:
Asthma function | 6 months
  Change in FEV1 (Forced expiratory volume in one second)

CONTACTS AND LOCATIONS:
Overall Officials: elena Curto, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided